CLINICAL TRIAL: NCT03649451
Title: Reference Dose Levels During Fluoroscopically Guided Procedures Performed Using Mobile X-ray Systems in Operating Rooms
Brief Title: Reference Dose Levels During Fluoroscopically Guided Procedures in Operating Rooms
Status: Completed | Type: Observational
Sponsor: Societe Francaise de Physique Medicale (Other)
Collaborators: Hopital Lariboisière (Other); University hospital, Angers, FRANCE (Unknown); University hospital of Montpellier, FRANCE (Unknown); Fréjus-Saint-Raphaël hospital, FRANCE (Unknown); C2i Santé, FRANCE (Unknown)
Responsible Party: Sponsor
Other Study IDs: gtsfpmnrbloc2017
Record Dates: First submitted 2018-08-02; First posted 2018-08-28 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Radiation Exposure
Keywords: Reference dose levels; Surgery; C-arm; Orthopedic; Urology; Vascular; Neurosurgery; Cardiology; Digestive; Fluoroscopy; Patient radiation protection; X-ray; Interventional radiology; Optimization; Kerma Area Product

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is conducted by a working group of the French Society of Medical Physics (SFPM). Its main aim is to establish reference dose levels for the most common procedures performed in operating rooms using mobile X-ray systems, hence helping medical physicists and surgeons to evaluate their practice and optimize patient radiation protection.

This is a multi-centric prospective study involving 73 medical institutions of different categories (public university hospitals, clinics, centers dedicated to cancer treatment, etc.). It consists on progressively collecting anonymous data for 15 to 30 procedures from a list of 62 types of procedures, belonging to 7 surgery specialties (neurosurgery, orthopedic surgery, digestive surgery, urology, cardiology, vascular surgery and multi-specialty). Collected data include patient BMI and information about the X-ray equipment, the medical procedure and the dosimetric parameters. Data collection doesn't require the access to the patient medical record and doesn't impact his medical care.

Proposed dose reference levels will be expressed in terms of KAP (Kerma-Area-Product), fluoroscopy time and air Kerma. Moreover, multiple statistical analyses will be done to investigate the impact of different variables on the procedure X-ray doses.

DETAILED DESCRIPTION:
Context:

Reference dose levels, introduced by the International Commission on Radiological Protection (ICRP) in 1996, are intended to help professionals using medical imaging to evaluate their practice and optimize patient's doses. European directive 2013/59/Euratom emphasizes the need to establish, use and regularly review reference levels for diagnostic and interventional procedures and to publish guidelines on this topic. Furthermore, national reference levels were established for conventional radiology and CT exams. They are used as a tool for the optimization of medical practices. Besides, a working group of the French Society of Medical Physics (SFPM) has published in 2017 reference levels for interventional radiology procedures performed in a dedicated room and using fixed angiographic equipment. Although radiation protection is a big challenge encountered in operating rooms using mobile X-ray equipment, few data are available in the literature regarding the use of this type of equipment.

In this context, the SFPM suggested the creation of a working group in 2017 to establish reference levels for the main procedures realized in the operating rooms using mobile X-ray systems. The aim of this working group is to help medical physicists and surgeons in evaluating their practice and optimizing patient radiation protection.

Scope of the study: The main purpose of the study is to establish dosimetric reference levels, in terms of KAP (Kerma-Area-Product). Additional objectives consist on proposing reference levels in terms of fluoroscopy time and air kerma and on studying the impact of different parameters (surgical specialty, body mass index, use of zoom, fluoroscopy pulse rate) on the delivered doses.

Study type and cohort: This is a multi-centric prospective study which consists on progressively collecting anonymous data for 15 to 30 procedures from a list of 62 surgical procedures (n=62) belonging to 7 different surgery specialties. Selected specialties are neurosurgery (n=12), orthopedic surgery (n=15), digestive surgery (n=6), urology (n=10), cardiology (n=6), vascular surgery (n=11), multi-specialty (n=2). 73 health institutions of different categories (University hospitals, clinics, centers dedicated to cancer treatment, etc..) confirmed their participations to the study.

Data collection: Data will be collected using a password-protected Excel spreadsheet. This excel file will be sent to all the participating institutions at the beginning of data collection. Every institution will send the excel file completed with anonymized data to the scientific responsible of the study through the secure email server of the APHP (Assistance Publique des Hopitaux de Paris)) institution.

Analysis: The main goal of this study is to publish descriptive statistics parameters (mean, standard deviation, median, 1st quartile, 3rd quartile) for each dosimetric data (KAP, fluoroscopy time, kerma, etc..) and for each category of surgical procedures. Results will be presented with a 95 percentage confidence interval.

Moreover, correlation analysis between several variables will be done. The differences between detector and equipment technologies will be also studied using appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Fluoroscopy guided procedures performed on adult patients (≥16 years old)
* Fluoroscopy guided procedures performed with mobile X-ray systems. Procedures performed outside of the operating rooms but using mobile X-ray systems are included in this study.
* Fluoroscopy guided procedures performed using mini C-arms or O-arms

Exclusion Criteria:

* Fluoroscopy guided procedures performed on pediatric patients (<16 years old)
* Fluoroscopy guided procedures performed with a fixed interventional radiology imaging system even if it was located in the operating rooms .
* Medical procedures performed using both a mobile X-ray system and a fixed CT scanner.
* Medical procedures performed using a mobile intra-operative CT scanner

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population consists on unhealthy patients undergoing surgical procedures with the use of X-ray mobile equipement. 62 types of procedures, belonging to 7 surgery specialties (neurosurgery, orthopedic, digestive, urology, cardiology, vascular and multi-specialty) are included in this study. For each procedure and each participating institution among the 73 centers that have sent their participation agreement, 15 to 30 procedures will be collected and analysed.
Sampling Method: Non-Probability Sample
Enrollment: 8840 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Total KAP (Kerma-Air-Product) | KAP is provided by the X-ray equipment at the end of the procedure.
  KAP or Kerma-Area-Product is the main dosimetric parameter representing the patient exposure. Participants should choose the appropriate unit of the KAP among a list of five units (microGray.m², milliGray.centimeter², centiGray.centimeter², deciGray.centimeter², Gray.centimeter²). Note that Gray is the international unit of the radiation quantity.

SECONDARY OUTCOMES:
Year of construction of the equipment and date of the last external quality control (QC) (yyyy) | baseline
  Year of construction of the equipment and date of the last external quality control
Image receptor type of the equipment | baseline
  Participants should specify whether the images are obtained using a flat panel detector or an X-ray image intensifier.
DACS Connection | baseline
  Participants should specify If the X-ray equipment is connected to a Dose Archiving and a Communication system (DACS) (Yes/no)
Patient weight (kg) and height (cm) | Patient weight and height are provided from the equipment or given by the medical team during the procedure
  Weight and height will be combined to report BMI in kg/m^2.
Size of Fields of View (FOV) (cm) | Baseline, The most used FOV during the procedure is provided by the medical staff
  Size of the smallest and largest Field of View (FOV); size of the largest FOV adapted to the size of the phantom; size of the most used FOV for the concerned procedure. (cm)
Differences between the displayed and measured X-ray doses (percentage) | baseline
  Differences between the displayed and measured KAP for the smallest and biggest FOV; Differences between the displayed and measured air kerma available in the last quality control (QC) report. (Percentages).
Total air kerma of the procedure including the one performed of an O-arm equipment | Data are provided by the X-ray equipment at the end of the procedure
  Participants should specify the unit by choosing the appropriate one among a list of 5 units (micro Gray, milli Gray, centi Gray, deci Gray, Gray).
Total number of image frames (number) | Data are provided by the X-ray equipment at the end of the procedure
  Total number of image frames (number)
Fluoroscopy mode used during the procedure | Data are provided by the X-ray equipment at the end of the procedure
  Participants should specify whether continuous, pulsed or mixed fluoroscopy modes are used during the procedure
Fluoroscopy pulse rate ( pulses/second) | Data are provided by the X-ray equipment at the end of the procedure
Fluoroscopy time (hh:mm:ss) of the procedure including the one performed of an O-arm equipment | Data are provided by the X-ray equipment at the end of the procedure
KAP (Kerma-Area-Product) attributable to fluoroscopy | Data are provided by the X-ray equipment at the end of the procedure
  Participants should choose the appropriate unit of the KAP among a list of five units (µGy.m², mGy.cm², cGy.cm², dGy.cm², Gy.cm²).
Medical specialty of the procedure | Data are provided by the medical staff during the procedure
  Participants should specify the medical specialty of the procedure by selecting one from a predefined list of seven categories: Orthopedic surgery, neurosurgery, cardiology, vascular surgery, urology, digestive surgery and multi-specialty.
Name/type of the procedure | Data are provided by the medical staff during the procedure
  Participants should specify the medical description of the procedure.
Additional information about the procedure giving further indications about the used materials or the anatomical region of interest. | Data are provided by the medical staff during the procedure
Total KAP for procedures performed on an O-arm equipment | KAP is provided by the X-ray equipment at the end of the procedure
  Participants should choose the appropriate unit of the KAP among a list of five units (µGy.m², mGy.cm², cGy.cm², dGy.cm², Gy.cm²).
Total DLP (Dose-Length-Product) of the procedures performed on an O-arm equipment.DLP is always expressed in mGy.cm. | DLP is provided by the X-ray equipment at the end of the procedure
  The DLP (Dose Length Product) is expressed in milliGray *centimeters (mGy.cm)
CTDIvol (Volume Computed Tomography Dose Index) of the procedures performed on an O-arm equipment. CTDI is always expressed in mGy. | CTDIvol is provided by the X-ray equipment at the end of the procedure
  The CTDIvol is a standardized measure of radiation dose output of a CT scanner. This dose is expressed in milliGrays (mGy).
Type of the dosimetric phantom used to calculate the CTDI of an acquisition for the procedures performed on an O-arm equipment. | Data are provided by the X-ray equipment at the end of the procedure
  Participants should select between a "head phantom (16 cm)" or a "body phantom (32 cm)"

CONTACTS AND LOCATIONS:
Overall Officials: Djamel DABLI, PhD, Principal Investigator — University hospital of Nîmes, France; Brice ROYER, MS, Principal Investigator — C2i Santé, FRANCE; Mathilde DEMONCHY, PhD, Principal Investigator — Fréjus-Saint-Raphaël hospital, FRANCE; Julien LE ROY, PhD, Principal Investigator — University hospital of Montpellier, FRANCE
Locations (1):
- Hopital Lariboisiere, Paris, France

IPD SHARING:
Plan to Share IPD: No
Only the final results of this study will be shared with the medical physicist members of the French Society of Medical Physicist. These results are statistical data analysis based on the collected patient data.
  Moreover, the study main results would be probably shared with the scientific community through a published paper in a scientific peer-reviewed journal.

DOCUMENTS (1):
  • Study Protocol (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT03649451/Prot_000.pdf